CLINICAL TRIAL: NCT01342744
Title: Effects of Metformin on Cardiovascular Risk Factors in Postmenopausal Women With Metabolic Syndrome
Brief Title: Metformin in Postmenopausal Women With Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Suchada Indhavivadhana, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si091/2011
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Metabolic Syndrome
Keywords: Cardiovascular risk factors
MeSH Terms: conditions — Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin (850mg) 1 tab oral twice a day
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo 1 tab oral twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin(850 mg) 1tab oral twice aday
  Arms: Metformin
Drug: Placebo — Placebo 1 tab oral twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of metformin on cardiovascular risk factors in postmenopausal women with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 45-60 years with metabolic syndrome according to The American Heart Association and The National Heart, Lung, and Blood Institute

Exclusion Criteria:

* Previous cardiovascular diseases
* Contraindicated to metformin: serum creatinine >1.4 mg/dL, liver disease, alcoholism, congestive heart failure, chronic hypoxic lung disease, prior history of lactic acidosis
* Previous administration of metformin, other hypoglycemic drugs, lipid-lowering drugs, sex steroids, antiplatelet drugs within 3 months before enrollment
* Fasting blood sugar ≥ 200 mg/dL or HbA1c >8%
* Serum triglyceride ≥500 mg/dL
* Abnormal EKG

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk factors | 6 months
  To compare the cardiovascular risk factors, including blood pressue, fasting blood sugar (FBS), Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR), 75-g oral glucose tolerance test (75-g OGTT), lipid profile, high sensitivity C-reactive protein(hs-CRP), neck circumference and waist circumference, between metformin and plcebo at 6 months

SECONDARY OUTCOMES:
10-year risk of coronary heart disease | 6 months
  To compare 10-year risk of coronary heart disease, which is calculated from RAMA- Electricity Generating Authority of Thailand (RAMA-EGAT) score, between metformin group and placebo at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suchada Indhavivadhana, M.D., Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand